CLINICAL TRIAL: NCT04938115
Title: Cell Therapy for CD7 Positive Acute Leukemia or Mixed Lineage Leukemia Except Those Who Are Diagnosed With T-ALL/T-LBL Using CD7-Specific CAR-T Cells
Brief Title: Cell Therapy for CD7 Positive Acute Myeloid Leukemia or Mixed Lineage Leukemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hebei Senlang Biotechnology Inc., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CD7+ mixed lineage leukemia
Record Dates: First submitted 2021-06-16; First posted 2021-06-24 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2023-05

CONDITIONS: Leukemia, T Cell
MeSH Terms: conditions — Leukemia, T-Cell

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CD7 CAR-T (Experimental)
  Interventions: Biological: CD7 CART

INTERVENTIONS:
Biological: CD7 CART — Biological: CD7 CAR-T; Drug: Cyclophosphamide,Fludarabine; Procedure: Leukapheresis

SUMMARY:
This is an open, single-arm, clinical study to evaluate efficacy and safety of anti CD7 CAR-T cell in the treatment of CD7 Positive acute leukemia or mixed lineage leukemia except those who are diagnosed with T-ALL/T-LBL

DETAILED DESCRIPTION:
The CARs consist of an anti-CD7 VHHs, a portion of the human CD137（4-1BB） molecule, and the intracellular component of the human CD3ζ molecule. Prior to CAR-T cell infusion, the patients will be subjected to preconditioning treatment. After CAR-T cell infusion, the patients will be evaluated for adverse reactions and efficacy.

The Main research objectives:

To evaluate the safety and efficacy of CD7 CAR-T cells in patients with CD7 Positive acute leukemia or mixed lineage leukemia except those who are diagnosed with T-ALL/T-LBL

The Secondary research objectives:

To investigate the cytokinetic characteristics of CD7 CAR-T cells in patients with CD7 Positive acute leukemia or mixed lineage leukemia except those who are diagnosed with T-ALL/T-LBL

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of refractory or relapsed CD7+ acute myeloid leukemia or mixed lineage leukemia was made according to the NCCN 2019.V2 guideline. Refractory AML is defined as a patient who has failed to achieve complete remission after induction therapy. Relapsed AML is defined as the reappearance of blasts (5%) in either peripheral blood or bone marrow. Patient diagnosed with AML should be treated and whose disease failed with at least 2 prior lines of therapies. Patients whose tumor burden ≥5% blasts, or who have persistent positive minimal residual disease (MRD), or have reappearance of extramedullary lesions are also considered eligible;
2. CD7+ expression on tumor cells (CD7 positive blasts ≥50% by flow cytometry);
3. Life expectancy greater than 12 weeks;
4. KPS or Lansky score≥60;
5. HGB≥70g/L (can be transfused);
6. oxygen saturation of blood>90%;
7. Total bilirubin (TBil)≤3 × upper limit normal, aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 5×upper limit of normal;
8. Informed consent explained to, understood by and signed by patient/guardian

Exclusion Criteria:

1. Any of the following cardiac criteria: Atrial fibrillation/flutter; Myocardial infarction within the last 12 months; Prolonged QT syndrome or secondary prolonged QT, per investigator discretion. Cardiac echocardiography with LVSF (left ventricular shortening fraction)<30% or LVEF(left ventricular ejection fraction)<50%; or clinically significant pericardial effusion. Cardiac dysfunction NYHA(New York Heart Association) III or IV (Confirmation of absence of these conditions on echocardiogram within 12 months of treatment);
2. Has an active GvHD;
3. Has a history of severe pulmonary function damaging;
4. With other tumors which is/are in advanced malignant and has/have systemic metastasis;
5. Severe or persistent infection that cannot be effectively controlled；
6. Merging severe autoimmune diseases or immunodeficiency disease;
7. Patients with active hepatitis B or hepatitis C([HBVDNA+]or [HCVRNA+]);
8. Patients with HIV infection or syphilis infection;
9. Has a history of serious allergies on Biological products (including antibiotics);
10. Clinically significant viral infection or uncontrolled viral reactivation of EBV(Epstein-Barr virus), CMV(cytomegalovirus), ADV(adenovirus), BK-virus, or HHV(human herpesvirus)-6;
11. Presence of symptomatic disorders of the central nervous system, which include but not limited to uncontrolled epilepsy, cerebrovascular ischemia/hemorrhage, dementia, and cerebellar disease, etc.;
12. Have received transplant treatment for less than 6 months in prior to enrollment;
13. Being pregnant and lactating or having pregnancy within 12 months;
14. Any situations that the researchers believe will increase the risks for the subject or affect the results of the study

Ages: 2 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-05-10 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-10-30 (Actual)

PRIMARY OUTCOMES:
Safety: Incidence and severity of adverse events | First 1 month post CAR-T cells infusion
  To evaluate the possible adverse events occurred within first one month after CD7 CAR-T infusion, including the incidence and severity of symptoms such as cytokine release syndrome and neurotoxicity
Efficacy: Remission Rate | 3 months post CAR-T cells infusion
  In the presence of extramedullary lesions, complete remission (CR), partial remission (PR), stable disease (SD), disease recurrence or progression (PD) shall be used to describe extramedullary lesions

SECONDARY OUTCOMES:
duration of response (DOR) | 24 months post CAR-T cells infusion
  duration of response (DOR)
Efficacy: progression-free survival (PFS) | 24 months post CAR-T cells infusion
  progression-free survival (PFS) time
CAR-T proliferation | 3 months post CAR-T cells infusion
  the copy number of CD7 CAR- T cells in the genomes of PBMC by qPCR method
CAR-T proliferation | 3 months post CAR-T cells infusion
  percentage of CD7 CAR- T cells measured by flow cytometry method
Cytokine release | First 1 month post CAR-T cells infusion
  Cytokine( IL-6,IL-10,IFN-γ,TNF-α ) concentration (pg/mL) by flow cytometry method
Pharmacokinetics (PK) indicators | 24 months post CAR-T cells infusion
  the peak concentration of Senl-T7 CAR-T cells amplified in the peripheral blood (Cmax, detected by flow cytometry and qPCR); the time taken to reach the peak concentration (Tmax), and the persistent time of the Senl-T7 CAR-T cells in vivo in patients
Pharmacodynamic (PD) indicators | First 1 month post CAR-T cells infusion
  the pharmacodynamic change in the clearance of peripheral blood CD7+ cells and the release of the cytokines at each observation time point

CONTACTS AND LOCATIONS:
Overall Officials: Peihua MD Lu, PhD, Principal Investigator — Hebei Yanda Ludaopei Hospital
Locations (1):
- He bei Yan da Lu dao pei Hospital, Beijingcun, Hebei, China

REFERENCES:
- [Derived] Lu P, Zhang X, Yang J, Li J, Qiu L, Gong M, Wang H, Chen J, Liu H, Xiong M, Liu Y, Wang L. Nanobody-based naturally selected CD7-targeted CAR-T therapy for acute myeloid leukemia. Blood. 2025 Mar 6;145(10):1022-1033. doi: 10.1182/blood.2024024861. PMID 39561281